CLINICAL TRIAL: NCT01424709
Title: Individualized 1st Line Chemotherapy Based on BRCA1 and RRM1 mRNA Expression Levels for Advanced Non-small Cell Lung Cancer
Brief Title: Individualized Chemotherapy Based on BRCA1 and RRM1 mRNA for Advanced Non-small Cell Lung Cancer (NSCLC)
Acronym: BRAVO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Caicun Zhou, Tonji University Affiliated Shanghai Pulmonary Hospital, Tongji University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRAVO study
Record Dates: First submitted 2011-05-09; First posted 2011-08-29 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Chemotherapy; Individual therapy; RRM1; BRCA1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Based on expression levels of RRM1 and BRCA1 mRNA，one of the four regimens will be given to each patient: Gemcitabine/cisplatin, Docetaxel/gemcitabine, CPT-11/Cisplatin, docetaxel monotherapy. The chemotherapy will be repeated every 3 week. Dose reduction or interruption for toxicity could take place at any time.
  Interventions: Drug: Gemcitabine, Docetaxel, CPT-11,Cisplatin
- Arm 2 (Active Comparator): gemcitabine/cisplatin up to 6 cycles or disease progression or intolerable toxicity.
  Interventions: Drug: gemcitabine/cisplatin

INTERVENTIONS:
Drug: Gemcitabine, Docetaxel, CPT-11,Cisplatin — Based on expression levels of RRM1 and BRCA1 mRNA，one of the four regimens will be given to each patient: Gemcitabine/cisplatin, Docetaxel/gemcitabine, CPT-11/Cisplatin, docetaxel monotherapy. The chemotherapy will be repeated every 3 week. Dose reduction or interruption for toxicity could take place at any time.
  Other Names: gemcitabine:Gemzar; Docetaxel:Taxotere; CPT-11:Irinotecan
  Arms: Arm 1
Drug: gemcitabine/cisplatin — gemcitabine/cisplatin up to 6 cycles or disease progression or intolerable toxicity.
  Other Names: gemcitabine:Gemzar
  Arms: Arm 2

SUMMARY:
Gemcitabine, docetaxel, CPT-11 and cisplatin are effective in 1st line treatment of advanced non-small cell lung cancer (NSCLC). Platinum-based doublets including gemcitabine, docetaxel or CPT-11 are standard 1st regimens. BRCA1 and RRM1 expression levels are reported to be associated with sensitivity of the tumor cells to cytotoxic agents. Some Phase II or III trials did prove feasibility of customized chemotherapy based upon expression levels of one or two biomarkers in the NSCLC patients. The investigators think customized chemotherapy may further improve efficacy of chemotherapy in advanced NSCLC. But there is no randomised trial to compare efficacy of standard chemotherapy with individualized chemotherapy in this setting. So, the investigators plan to initiate this phase II trial to compare efficacy between standard chemotherapy of gemcitabine/cisplatin versus customized chemotherapy in chemonaive NSCLC patients.

DETAILED DESCRIPTION:
Primary end point:ORR Secondary end point:PFS,OS,safety,QOL,etc.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent,
2. Histologically confirmed stage M1a or M1b NSCLC,
3. Aged over 18 years old,
4. Measurable disease,
5. Life expectancy of at least 12 weeks,
6. No prior chemotherapy or target therapy,
7. No brain metastases or spinal cord compression,
8. Less than 10% body weight loss,
9. ECOG performance status 0-2,
10. Adequate vital organ function (haematological, renal, hepatic, etc).
11. Enough tissue for detection of BRCA1 and RRM1 expression.

Exclusion Criteria:

1. Prior systemic cytotoxic chemotherapy or EGFR TKI therapy,
2. Positive pregnancy test,
3. Another active malignancy, other than superficial basal cell and squamous cell or carcinoma in situ of the cervix, within the last 5 years,
4. Patients with brain metastases or spinal cord compression,
5. Allergy to gemcitabine, cisplatin, docetaxel, CPT-11,
6. Any unstable systemic disease including active infection,
7. No enough tissue for detection of BRCA1 and RRM1

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-12; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | tumor assessment 6-8 weeks after the initiation of chemotherapy
  to evaluate ORR during 6-8 weeks after all cycles complete

SECONDARY OUTCOMES:
Progression free survival | 24 months
  PFS is evaluated in the 24th month since the treatment began
duration of response | 24 months
  evaluated in the 24th month since the treatment began
overall survival | 24 months
  evaluated in the 24th month since the treatment began
safety | 24 months
  evaluated in the 24th month since the treatment began
Quality Of Life | 24 months
  evaluated in the 24th month since the treatment began

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Ph.D, Principal Investigator — Tongji University Affiliated Shanghai Pulmonary Hospital
Locations (1):
- Medical Department, Shanghai Pulmonary Hospital, Shanghai, China